CLINICAL TRIAL: NCT02352441
Title: Cognitive Rehabilitation:ACTION Training for Soldiers With Executive Dysfunction
Acronym: ACTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Mary Radomski, Senior Scientific Advisor, Allina Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11215006
Record Dates: First submitted 2015-01-23; First posted 2015-02-02 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implementation Intentions (Experimental): This group will receive training in Implementation Intentions during 3 sessions, 1 day/week, over 3 weeks. They will receive usual care through the standard program, 1 day/week during these 3 weeks.
  Interventions: Other: Implementation Intentions(II)
- Usual Care (No Intervention): This group will participate in the usual group intervention provided to Service members experiencing executive dysfunction associated with mild traumatic brain injury, 2 days / week during 3 weeks.

INTERVENTIONS:
Other: Implementation Intentions(II) — Implementation Intention training will include:
  Demonstration and practice using examples and personal goals identified at first session. Worksheets will be provided to practice IF-THEN statements to set Implementation Intentions. Additionally, at the end of each session, the participant will be instructed to perform and event based or time based task. The objective is to see if those receiving II training are more likely to carry out the assigned task than those who do not receive II training. They will also be expected to practice II at least 5 days/week using personal goals.
  Arms: Implementation Intentions

SUMMARY:
Many Service members (SM) experience executive dysfunction associated with mild traumatic brain injury symptom complex (mTBI-sc), for which they receive cognitive rehabilitation. Cognitive rehabilitation (CR) for executive dysfunction often involves metacognitive strategy instruction (MSI) to help patients self-regulate their behavior though a goal management process - identifying a goal, anticipating performance problems, generating possible solutions, self-monitoring performance during the activity, recognizing maladaptive task strategies, stopping and then modifying real-time task behavior by choosing an alternate strategy. MSI alone often does not result in improved daily functioning because it requires conscious cognitive oversight to employ (which is difficult for people with executive dysfunction) and it presumes that simply establishing goals propels goal-directed action, when for many people, this is not so. Social psychologists report that people who set implementation intentions (if-then statements that link specific situational cues with specific goal actions) are more likely to perform goal actions than those who only set goal intentions. Implementation intentions are believed to be effective because they enable people to switch from conscious-effortful reflective action control to automatic, reflexive action control associated with selected situational cues. A team of researchers from the Courage Kenny Research Center (CKRC), Traumatic Brain Injury Center at Fort Campbell, KY (TBIC-FC), and Neurofunctional Research and Consulting has developed a brief CR intervention to teach SM with mTBI-sc to set implementation intentions called ACTION (AutomatiC iniTiation of IntentiONs) sequence training. The purpose of this pilot study to evaluate: 1) the practicality of instructional methods used to teach SM with mTBI-sc to perform the ACTION sequence and 2) the efficacy of ACTION sequence training in achieving personal goals and performance on a task that challenges executive function using a small randomized controlled trial. If the results are positive, a larger study would be conducted to determine the impact of ACTION sequence training on SM performance on military-relevant tasks and goals.

DETAILED DESCRIPTION:
The primary aims of this feasibility study are as follows:

Aim 1: Finalize ACTION training curriculum; develop manuals; field test .

* Work with implementation intentions research expert and a military consultant to develop a training task gradation schema which informs the identification and modification of existing implementation intentions training tasks so that they have military face validity.
* Finalize the adherence support methods and other training worksheets and materials.
* Field test training tasks and adherence support methods on small cohort of civilians with mTBI-sc from CKRC to assure feasibility.
* Finalize ACTION sequence training manuals; assure intra-rater and inter-rater reliability for scoring quality of implementation intentions statements.

Aim 2: Evaluate ACTION sequence training instructional methods (the extent to which SM with mTBI-sc are able to learn to establish IF-THEN statements that have the potential to trigger automatic enactment of goal-actions and the extent to which SM with mTBI-sc report the training experience as satisfactory and beneficial).

* Enroll up to 28 participants in the study (SM with mTBI-sc who are referred to MSI at TBIC-FC).
* Evaluate whether or not participants can correctly craft implementation intentions by using a rubric to score implementation intentions developed by participants during clinic sessions and during home practice; administer participation satisfaction survey at posttest.

Aim 3: Test the efficacy of ACTION sequence training by evaluating the extent to which training 1) improves SM's with mTBI-sc ability to perform a complex test of executive function (e.g. Hotel Test) and 2) advances progress towards self-identified goals in daily life (via Canadian Occupational Performance measure [COPM] and Goal Attainment Scaling [GAS]) as compared to a control condition. Additionally, determine level of adherence to completing daily homework practice ans assigned prospective memory tasks.

* Collect pre-post data on the Hotel Test, COPM, GAS on all participants.
* Collect data on completion of homework assignments
* Collect data on completion of prospective memory tasks

ELIGIBILITY:
Inclusion Criteria:The sample population at the Traumatic Brain Injury Clinic- Fort Campbell (TBIC-FC) will consist of active duty army soldiers, reservists, national guardsmen, airmen, and retirees; the majority of the sample population will be active duty army soldiers. Study volunteers will be recruited from among service members assessed in the TBIC-FC and referred to the Cognitive Clinic for performance problems secondary to reported / suspected combat-related mTBI-sc.

-

Exclusion Criteria:Not willing to sign consent to participate.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change in performance of the Hotel Task | Baseline and end of 3 weeks
  The Hotel Task requires the participant to perform a set of 6 tasks in 10 minutes with the instruction to perform all tasks with no expectation for completing any of the tasks. This task tests the ability of the participant to shift. Measurements associated with this task include time spent on each task and number of tasks completed.
Change in the Canadian Occupational Performance Measure | Baseline and end of 3 weeks
  Participants will provide their self-perceived performance on three everyday tasks identified and prioritized as problematic.
Change in Goal Attainment Scaling | Baseline and end of 3 weeks
  Attainment of five goals linked to selected five everyday tasks

SECONDARY OUTCOMES:
Performance of assigned tasks given at the end of each of the 6 II sessions | End of sessions 1 and 2 for each of weeks 1, 2, and 3
  Monitoring performance of the assigned event or time based task, Yes(2 points)/No(0 points)/Partial(1 point)
Performance of homework | 4 days / week for each of the 3 weeks of study participation
  Participant will be expected to call in and report having done assignment

CONTACTS AND LOCATIONS:
Overall Officials: Mary Radomski, OTR/L, PhD, Principal Investigator — Allina Health; Mark Showers, MS, OTR/L, Principal Investigator — Fort Campbell
Locations (1):
- Fort Campbell Intrepid Spirit, Fort Campbell North, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radomski MV, Giles GM, Owens J, Showers M, Rabusch S, Kreiger R, Zola J, Kath K. Can service members with mild traumatic brain injury learn to develop implementation intentions for self-identified goals? Disabil Rehabil. 2022 Jun;44(12):2640-2647. doi: 10.1080/09638288.2020.1841309. Epub 2020 Nov 4. PMID 33147426